CLINICAL TRIAL: NCT06439589
Title: An Open-label, Multi-center Phase Ib/II Study of HRS2398 in Combination With Adebrelimab in Patients With Advanced Solid Tumors
Brief Title: Phase Ib/II Study of HRS2398 in Combination With Adebrelimab in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS2398-201-PD-L1
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS2398 given in combination with adebrelimab (Experimental)
  Interventions: Drug: HRS2398; Drug: Adebrelimab

INTERVENTIONS:
Drug: HRS2398 — HRS2398: Tablets, 40mg/tablet, oral
Drug: Adebrelimab — Adebrelimab (SHR-1316): injection, 600mg(12mL), intravenous infusion

SUMMARY:
This study is a multicenter, open-label, dose-finding/efficacy-expanding phase Ib/II clinical trial, which aims to observe and evaluate the tolerability, safety, pharmacokinetic characteristics and immunogenicity of HRS2398 combined with Adebrelimab injection in patients with advanced solid tumors, determine the RP2D, and preliminarily evaluate the efficacy of HRS2398 combined with Adebrelimab in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are able to give voluntary informed consent, understand the study and are willing to follow and complete all the test procedures.
2. Age 18~75 years old.
3. Dose escalation phase: patients with clinically diagnosed or pathologically confirmed advanced solid tumors who have failed standard therapy (disease progression during or after treatment) or for whom no effective standard treatment regimen exists.
4. Dose Expansion and Efficacy Expansion Phase: Patients with advanced solid tumors who have received systemic immunotherapy and platinum-containing chemotherapy in the recurrent/metastatic settings.
5. At least one measurable lesion per RECIST v1.1 criteria.
6. ECOG PS score: 0-1.

Exclusion Criteria:

1. Patients with meningeal metastases; or with brain metastases that have not been treated with surgery or radiotherapy.
2. Cancerous ascites and pleural effusion with clinical symptoms, requiring puncture and drainage; or those who have received ascites, pleural effusion drainage within 14 days before the first dose.
3. Presence of any active, known autoimmune disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The number of subjects with dose-limiting toxicity (DLT) | From first dose of study treatment until the end of Cycle 1（up to 28 days）
Determination of Recommended Phase II dose (RP2D) | From first dose of study treatment until the end of Cycle 1（up to 28 days）
Objective Response Rate (ORR) | From time of first dose of HRS2398 or Adebrelimab until the date of objective disease progression or death (up to 6 months)

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | From time of first dose of HRS2398 or Adebrelimab until the date of objective disease progression or death (up to 6 months)
Duration of Response (DoR) | From time of first dose of objective disease progression until the date of objective disease progression or death (up to 6 months)
Progression free Survival (PFS) | From time of first dose of objective disease progression until the date of objective disease progression or death (up to 6 months)
Overall Survival (OS) | From time of first dose of objective disease progression until the date of death (up to 24 months)
Time To Response(TTR) | From time of first dose of objective disease progression until the date of objective disease progression or death (up to 6 months)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided